CLINICAL TRIAL: NCT02954822
Title: A Randomized, Open-label, Multiple Dosing, Cross-over Clinical Trial to Investigate the Pharmacokinetic/Pharmacodynamic Drug-drug Interaction of Evogliptin 5mg and Glimepiride 4mg After Oral Administration in Healthy Male Subjects
Brief Title: Pharmacokinetic/Pharmacodynamic Drug-drug Interaction of Evogliptin 5mg and Glimepiride 4mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: DA1229_DIG_I
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- (Group A) (Experimental): Evogliptin→Evogliptin+Glimepiride→Glimepiride
  Interventions: Drug: Evogliptin→Evogliptin+Glimepiride→Glimepiride
- (Group B) (Experimental): Glimepiride→Evogliptin→Evogliptin+Glimepiride
  Interventions: Drug: Glimepiride→Evogliptin→Evogliptin+Glimepiride

INTERVENTIONS:
Drug: Evogliptin→Evogliptin+Glimepiride→Glimepiride — Evogliptin 5mg will be administered for 7days and then glimepiride 4mg will be added on and administered with Evogliptin 5mg for 2 days. After the washout period for 10 days, Glimepiride 4mg will be administered for 2 days.
  Glimepiride : Glimepiride 4mg QD
  Evogliptin + Glimepiride : Evogliptin 5mg QD + Glimepiride 4mg QD
  Other Names: Suganon, Amaryl
  Arms: (Group A)
Drug: Glimepiride→Evogliptin→Evogliptin+Glimepiride — After 2 days of administration of Glimepiride 4mg follows the 10-day washout period. Afterwards Evogliptin 5mg will be administered for 7days and then glimepiride 4mg will be added on and administered with Evogliptin 5mg for 2 days.
  Other Names: Suganon, Amaryl
  Arms: (Group B)

SUMMARY:
A randomized, open-label, multiple dosing, three treatment, three period, two sequence clinical trial to investigate the pharmacokinetic/pharmacodynamic drug-drug interaction of evogliptin 5 mg and glimepiride 4 mg after oral administration in healthy male subjects

DETAILED DESCRIPTION:
A randomized, open-label, multiple-dose, three-treatment, three-period, two-sequence, crossover study

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male Volunteers (Age: 19~45years)
* 55<Body Weight<90, 18<BMI<27
* FPG: 70-125 mg/dL

Exclusion Criteria:

* galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Clinically significant Medical History
* Allergy or Drug Hypersensitivity
* AST(SGOT), ALT(SGPT) > Upper Normal Range*1.5, eGFR<80 mL/min
* Drink during clinical trial period
* Smoking during clinical trial period
* Grapefruit/Caffeine intake during clinical trial period
* No Contraception

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss for Evogliptin and Glimepiride | 3 weeks
  area under the concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., Principal Investigator — Clinical Trial Center, Seoul National University Hospital
Locations (1):
- Clinical Trials Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided